CLINICAL TRIAL: NCT01695421
Title: Soft-hard Technologies to Assistance and Accessibility in Patients With Chronic Diseases: The Effect of a Five Week Electrical Myostimulation Program.
Brief Title: The Effect of a Five Week Electrical Myostimulation Program in Chronic Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Gerson Cipriano Jr, Professor, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CSF-01
Record Dates: First submitted 2012-09-19; First posted 2012-09-28 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2012-09

CONDITIONS: Heart Failure
Keywords: Transcutaneous Electric Nerve Stimulation; Oxygen Consumption; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Functional electrical stimulation (Experimental): Burst modulated alternating rectified current with a 10 Hz carrier frequency, 400 microsecond pulse duration and 50 Hz bursts
  Interventions: Procedure: Functional electrical stimulation
- Medium-frequency alternating current (Experimental): Burst modulated alternating current with a 2500 Hz carrier frequency, 400 microsecond pulse duration and 50 Hz bursts
  Interventions: Procedure: Medium-frequency alternating current
- Burst-modulated alternating current (Experimental): Burst modulated alternating current with a 4000 Hz carrier frequency, 400 microsecond pulse duration and 50 Hz bursts.
  Interventions: Procedure: Burst-modulated alternating current
- Placebo (Placebo Comparator): Training with the intensity of 5 mA.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Medium-frequency alternating current — The subjects will receive stimulation to quadriceps and gastrocnemius for 5 days a week for 1 hour during 5 weeks. Electrical stimulation will be delivered through channel one with one electrode placed over the vastus medialis and the second electrode placed medial and distal to the greater trochanter. The channel two will be place on the gastrocnemius with one electrode positioned over the muscle belly and the second over the musculotendinous junction. The stimulus will be on for 10 seconds followed by a 30 second relaxation period at the first two weeks. Subsequently, the EMS stimulus will be on for 15 seconds followed by a 30 second relaxation period. The intensity will be turned up to the maximal tolerable intensity as reported by the subject (10-100 mA) observing muscular contraction.
  Other Names: MAC
  Arms: Medium-frequency alternating current
Procedure: Burst-modulated alternating current — The subjects will receive stimulation to quadriceps and gastrocnemius for 5 days a week for 1 hour during 5 weeks. Electrical stimulation will be delivered through channel one with one electrode placed over the vastus medialis and the second electrode placed medial and distal to the greater trochanter. The channel two will be place on the gastrocnemius with one electrode positioned over the muscle belly and the second over the musculotendinous junction. The stimulus will be on for 10 seconds followed by a 30 second relaxation period at the first two weeks. Subsequently, the EMS stimulus will be on for 15 seconds followed by a 30 second relaxation period. The intensity will be turned up to the maximal tolerable intensity as reported by the subject (10-100 mA) observing muscular contraction.
  Other Names: BMAC
  Arms: Burst-modulated alternating current
Procedure: Placebo — The subjects will receive stimulation to quadriceps and gastrocnemius for 5 days a week for 1 hour during 5 weeks. Electrical stimulation will be delivered through channel one with one electrode placed over the vastus medialis and the second electrode placed medial and distal to the greater trochanter. The channel two will be place on the gastrocnemius with one electrode positioned over the muscle belly and the second over the musculotendinous junction. The stimulus will be on for 10 seconds followed by a 30 second relaxation period at the first two weeks. Subsequently, the EMS stimulus will be on for 15 seconds followed by a 30 second relaxation period. The intensity will be fixed on 5 mA.
  Arms: Placebo
Procedure: Functional electrical stimulation — The subjects will receive stimulation to quadriceps and gastrocnemius for 5 days a week for 1 hour during 5 weeks. Electrical stimulation will be delivered through channel one with one electrode placed over the vastus medialis and the second electrode placed medial and distal to the greater trochanter. The channel two will be place on the gastrocnemius with one electrode positioned over the muscle belly and the second over the musculotendinous junction. The stimulus will be on for 10 seconds followed by a 30 second relaxation period at the first two weeks. Subsequently, the EMS stimulus will be on for 15 seconds followed by a 30 second relaxation period. The intensity will be turned up to the maximal tolerable intensity as reported by the subject (10-100 mA) observing muscular contraction
  Arms: Functional electrical stimulation

SUMMARY:
Patients afflicted with Chronic Heart Failure (HF) typically do not maintain stable cardiac function for the remainder of their life and consequently require continuous medical management and intermittent hospital admissions. Several investigations have demonstrated that electrical muscle stimulation (EMS) produces positive physiologic and psychological adaptations in patients with HF. However not all the EMS modalities were been evaluated on this population or not even were tested based on present recognized gold standard clinical parameters after a short period of treatment. The primary aims of the proposed study is to: Determine the effect of a five week home based of three EMS modalities on prognostics markers, perceived quality of life, muscle force and electrical activity in subjects diagnosed with HF.

DETAILED DESCRIPTION:
Introduction: Chronic Heart Failure (HF) patients are a significant health care burden in many countries. Patients afflicted with HF typically do not maintain stable cardiac function for the remainder of their life and consequently require continuous medical management and intermittent hospital admissions. Several investigations have demonstrated that electrical muscle stimulation (EMS) produces positive physiologic and psychological adaptations in patients with HF. However not all the EMS modalities were been evaluated on this population or not even were tested based on present recognized gold standard clinical parameters after a short period of treatment. The impact of use of low frequency (FES) and medium-frequency currents (MAC and BMAC) as EMS on the VE/VCO2 and BNP has likewise not been investigated in patients with HF.

Purposes: The primary aims of the proposed study is to: Determine the effect of a five week home based EMS modalities (a) Functional electrical stimulation (FES), (b) medium-frequency alternating current (MAC) and (c) burst-modulated medium-frequency alternating current (BMAC) training program on the VE/VCO2 slope, Brain Natriuretic Peptide (BNP) level, peak VO2, VO2 at Ventilatory Threshold (VT), perceived quality of life, muscle force and electrical activity in subjects diagnosed with HF (NYHA III and IV). Examine changes in the previously outlined outcome measurements five weeks after cessation of the EMS ((a) FES, (b) MAC and (c) BMAC) training program.

Procedures: We will recruit 40 persons (10 for each EMS modalities and 10 control subjects) diagnosed with HF. A group of control subjects will participate using a sham current. The protocol can be conceptually divided into four sections in the following chronological sequence: (1) baseline assessment (body composition by a bone densitometer X-ray Dual energy X-Ray absortometry - DXA, Resting blood pressure and heart rate, complete blood count and BNP analysis); Living with Heart Failure Questionnaire (MLWHFQ); A physician-supervised maximal aerobic exercise test using a metabolic cart (Vmax, Viasys, USA) (VO2, VE/VCO2, VT); isokinetic peak torque (Biodex System III, Isokinetic Dynamometer, Biodex Medical, Inc., Shirley, NY) and electrical activity (Miotec, Brazil), (2) five week EMS training program (bilateral quadriceps and gastrocnemius for 5 days a week for 1 hour to each muscle group with FES, MAC and BMAC training program), (3) immediate post-training assessment within 5 days of completion of the EMS training program and a (4) final analysis five weeks after cessation of the EMS training program.

ELIGIBILITY:
Inclusion Criteria:

* (1) Male or female ≥ 21 and ≤ 80 years of age.
* (2) Current HF symptoms consistent with NYHA class III-IV.
* (3) On stable HF pharmacological therapy for at least one month prior to data collection.
* (4) Left ventricular ejection fraction < 45% documented within 3 months of enrollment (obtained from subjects medical records).
* (5) No planned elective surgery or pacemaker implantation at the time of study initiation.
* (6) Hgb > 8.0 within 1 month of enrollment (obtained from subjects medical records).
* (7) Willingness to provide written informed consent.

Exclusion Criteria:

* (1) Inability to provide written informed consent.
* (2) Inability to walk on a treadmill.
* (3) Hemodynamically significant valvular heart disease.
* (4) Unstable angina.
* (5) Acute myocardial infarction within the previous 3 months.
* (6) Obstructive hypertrophic cardiomyopathy.
* (7) HF known to be secondary to pericardial disease or uncorrected valvular disease.
* (8) Chronic oxygen therapy.
* (9) Participation in another clinical trial within the past 30 days.
* (10) Participation in a regular exercise within the previous 6 months.
* (11) Previous implantation of a cardiac pacemaker or defibrillator.
* (12) Pregnancy.
* (13) Resting systolic blood pressure > 200 mmHg.
* (14) Failure to demonstrate the ability to operate the EMS unit.
* (15) Failure to be compliant with at least 75% of the EMS training sessions.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
VE/VCO2 slope | Change from Baseline in VE/VCO2 slope at five and ten weeks post EMS.

SECONDARY OUTCOMES:
Peak VO2 | Change from Baseline in Peak VO2 at five and ten weeks post EMS.
VO2 at Ventilatory Threshold | Change from Baseline in VO2 at ventilatory threshold at five and ten weeks post EMS.
Perceived quality of life | Change from Baseline in perceived quality od life at five and ten weeks post EMS.
Muscle force | Change from Baseline in muscle force at five and ten weeks post EMS.
Muscle electrical activity | Change from Baseline in muscle electrical activity at five and ten weeks post EMS.
Brain Natriuretic Peptide level | Change from Baseline in Brain Natriuretic Peptide Level at five and ten weeks post EMS.

CONTACTS AND LOCATIONS:
Overall Officials: Gerson Cipriano Junior, PhD, Principal Investigator — University of Brasilia
Locations (1):
- Brasilia University, Brasília, Federal District, Brazil

REFERENCES:
- [Background] Myers J, Gademan M, Brunner K, Kottman W, Boesch C, Dubach P. Effects of high-intensity training on indices of ventilatory efficiency in chronic heart failure. J Cardiopulm Rehabil Prev. 2012 Jan-Feb;32(1):9-16. doi: 10.1097/HCR.0b013e3182343bdf. PMID 22113369
- [Background] Arena R, Myers J, Aslam SS, Varughese EB, Peberdy MA. Peak VO2 and VE/VCO2 slope in patients with heart failure: a prognostic comparison. Am Heart J. 2004 Feb;147(2):354-60. doi: 10.1016/j.ahj.2003.07.014. PMID 14760336
- [Background] Mueller C, Scholer A, Laule-Kilian K, Martina B, Schindler C, Buser P, Pfisterer M, Perruchoud AP. Use of B-type natriuretic peptide in the evaluation and management of acute dyspnea. N Engl J Med. 2004 Feb 12;350(7):647-54. doi: 10.1056/NEJMoa031681. PMID 14960741
- [Derived] Vieira PJ, Chiappa AM, Cipriano G Jr, Umpierre D, Arena R, Chiappa GR. Neuromuscular electrical stimulation improves clinical and physiological function in COPD patients. Respir Med. 2014 Apr;108(4):609-20. doi: 10.1016/j.rmed.2013.12.013. Epub 2014 Jan 2. PMID 24418570